CLINICAL TRIAL: NCT05953805
Title: Patients' and Healthcare Professionals' Experience of Using Apple iPads to Conduct Patient and Public Involvement Activity - a Qualitative Study
Brief Title: Exploring Patient and Staff Experience of Using iPads for PPI Activity
Acronym: LEAP
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19RM008
Record Dates: First submitted 2021-03-24; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients With iPads: Patients who have been assigned an iPad to complete their PPI sessions remotely
- Patients Without iPads: Patients who will continue to attend the classic face to face PPI meetings
- Staff: Staff who will give their opinions on the use of iPads against normal PPI methods

SUMMARY:
Patients' and healthcare professionals' experience of using Apple iPads to conduct patient and public involvement activity

DETAILED DESCRIPTION:
There is a long overdue push to get patients engaged at the earliest stage possible of the research cycle so there is earlier collaboration between the public/patients and the researcher rather than much later on in the research process. For this reason there are successful patient and public meetings that occur in various specialities within the NHS. However, attending these meetings can be difficult as timings for multiple people to attend at the same physical location can be logistically difficult. It can be further compounded if potential members are unable to attend due to their illness. For example, patients may be on home oxygen and therefore may not be selected by the facilitator or perhaps they themselves may decide to exclude themselves.

Previous research has had an online forum to engage the public/patients with the research process. However, the findings were that there was room to improve from an engagement perspective and furthermore, the real-time communication was limited due to how forums functions.

For this reason, the investigators have suggested using iPads so the investigators can have virtual meetings which negates the need to attend meetings physically. The investigators have used iPads instead of other tablets due to their higher encryption standards and because the in-built FaceTime is easier to use than other systems that install a separate application. Virtual meetings where a group of people are not in the same physical location and are communicating via telephone or the internet. Many patients who may not have been considered/been approached about being part of PPI can now participate virtually. In addition, the time commitment is significantly reduced as it would only involve the time the meeting would be held and not the travel time, which can be extensive.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* Part of a respiratory medicine PPI group or a PPI group that will be started prior to consent into the study at Nottingham University Hospital Trust

Exclusion Criteria:

* Adults lacking mental capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Participants in the PPI group and allocated an iPad: focus groups will be conducted either on hospital site or remotely using iPads.
  * Participants in PPI and not allocated an iPad: focus groups will be conducted on NUH premises.
  * Healthcare professionals involved in PPI activity with participants using iPad: docus group will be conducted at NUH
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Use of technology to perform remote PPI | Up to 12months
  To explore the patient and staff experience of using iPads for PPI sessions instead of physically attending meetings. Focus groups were used and were analysed using the DeLone model of information systems as the theoretical framework.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom